CLINICAL TRIAL: NCT03766373
Title: Evaluation of Safety and Reduction of Ear Pain in Adults With Acute Otitis Media
Brief Title: Evaluation of Safety and Reduction of Ear Pain in Adults With Acute Otitis Media and Reduction of Ear Pain in Adults With Acute Otitis Media
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novus Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: OP0201-C-004
Record Dates: First submitted 2018-12-03; First posted 2018-12-06 (Actual); Results first posted 2019-11-21 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-10

CONDITIONS: Acute Otitis Media
MeSH Terms: conditions — Otitis Media

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Drug: OP0201 (Active Comparator)
  Interventions: Combination Product: Drug: OP0201 20mg
- Drug: Placebo (Placebo Comparator)
  Interventions: Combination Product: Drug: Placebo 0mg

INTERVENTIONS:
Combination Product: Drug: OP0201 20mg — OP0201
  Arms: Drug: OP0201
Combination Product: Drug: Placebo 0mg — Placebo
  Arms: Drug: Placebo

SUMMARY:
The purpose of this study is to evaluate the Safety and Reduction of Ear Pain in Adults with Acute Otitis Media.

ELIGIBILITY:
Inclusion Criteria includes but is not limited to:

1. AOM diagnosis with moderate to severe bulging of the TM and recent (< 48 hours [h]) onset of ear pain.
2. Moderate to severe ear pain in the affected ear(s), defined as a score of ≥ 5 (on a scale of 0 10) on the NRS 11 as evaluated by the subject at Screening.
3. Generally good health (other than AOM) as determined by evaluation of medical history and physical examination at Screening.
4. Negative urine pregnancy test at Screening for all female subjects of childbearing potential.
5. Able to read and sign written informed consent prior to study participation.

Exclusion Criteria includes but is not limited to:

1. Presence of a perforated TM at Screening or had a perforated TM within 6 months (mo) prior to Screening as determined by medical history
2. Subjects with tympanostomy tubes
3. Acute or chronic otitis externa
4. Chronic otitis media defined as confirmed presence of middle ear effusion for 12 weeks or longer
5. Disorders with decreased mucociliary clearance or higher viscosity of the mucous (eg, cystic fibrosis, primary ciliary dyskinesia, Kartagener's syndrome)
6. Clinically relevant blockage of 1 or both nasal passages, as determined by the investigator's medical judgment
7. Permanent hearing loss irrespective of otitis media
8. Subjects with medical conditions that may affect interpretation of the safety or efficacy of study drug as determined by the investigator's medical judgment
9. Subjects with craniofacial abnormalities (eg, cleft palate, Down's Syndrome)
10. Subjects with erythema of the TM without other evidence of otitis media
11. Seborrheic dermatitis involving the affected external ear canal or pinna
12. Use of medications with known vasoconstrictive properties (eg, decongestants [Afrin®, Sudafed®]) currently or within 2 h prior to Screening
13. Use of oral analgesics < 2 h prior to Screening or Baseline (oral analgesics > 2 h are permitted as long as ear pain criteria are met per Inclusion Criteria)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-01-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - US Clinical Research Group, LLC., Bellflower, California
  - Vista Health Research, Miami, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://novustherapeutics.com/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Drug: OP0201 | Drug: Placebo
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Drug: OP0201 | Drug: Placebo | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (13.24) | 45.7 (16.15) | 49.5 (14.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 16
  Male | 2 | 6 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 7 | 16
  Not Hispanic or Latino | 3 | 5 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 1 | 2
  White | 9 | 7 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Time Frame: 1 Day
Measure: Count of Participants; unit: Participants
Arm/Group | Drug: OP0201 | Drug: Placebo
Number analyzed (Participants) | 12 | 12
Participants | 2 | 6

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Drug: OP0201 | Drug: Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 2/12 | 6/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug: OP0201 (N=12) | Drug: Placebo (N=12)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0)
Feeling cold (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-03-12): https://cdn.clinicaltrials.gov/large-docs/73/NCT03766373/SAP_000.pdf
  • Study Protocol (2018-07-10): https://cdn.clinicaltrials.gov/large-docs/73/NCT03766373/Prot_001.pdf